CLINICAL TRIAL: NCT04750876
Title: Early Evaluation of the Introduction of Pre- and Post-operative Psychological and Physiotherapeutic Follow-up in Vascular Surgery in Amputee Patients
Acronym: EPKIVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHD20_0056
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-07

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional support (Active Comparator)
  Interventions: Other: Conventional support
- Specific care, including the intervention of a psychologist and a physical therapist. (Experimental)
  Interventions: Other: Specific care, including the intervention of a psychologist and a physical therapist.

INTERVENTIONS:
Other: Conventional support — Patients in the "Conventional support" randomisation arm will follow the usual care of amputee patients in the vascular surgery department. They will be cared for by the surgeon, nurses and nursing auxiliaries, who will provide individualised care (nursing care, mobilisation, pain management, technical care, etc.), listening and support.
  Arms: Conventional support
Other: Specific care, including the intervention of a psychologist and a physical therapist. — In the case where the patient is in the "Specific care, including the intervention of a psychologist and a physical therapist." arm, the usual care will be associated with :
  * consultations with a psychologist
  * The patient will also be cared for on a daily basis by a physical therapist.
  Arms: Specific care, including the intervention of a psychologist and a physical therapist.

SUMMARY:
An amputation represents a real ordeal for the person who will have to overcome the loss of a limb and face long months of rehabilitation. It is most often carried out following arterial insufficiency.

As paramedical professionals, we see in our daily practice a physical and psychological suffering for amputee patients. In spite of our skills acquired through training and professional experience, we are unable to offer comprehensive care for these patients and therefore feel that we are offering incomplete care. A multidisciplinary care, including a medical and paramedical team, would seem to us to be more appropriate for patients with lower limb amputations.

Following this observation, we would like to highlight the interest for the patient and the care team to include a psychologist and a physiotherapist in the care offer to evaluate the improvement of the physical and emotional state of the amputee patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of majority, no age limit
* Amputation related to obliterative arteriopathy of the lower limbs
* Trans-tibial or trans-femoral amputation in an already amputated patient
* Patient with an indication of discharge to a rehabilitation and re-education service
* Patient with the ability to understand the protocol
* Patient who has agreed to participate in the study and has given express oral consent
* Patient receiving social security cover or entitled to it

Exclusion Criteria:

* Trauma related amputation
* Patient with no history of amputation
* Amputation of upper limb, trans-metatarsal or one or more toes
* Amputation of comfort in a palliative care setting
* Patient leaving home after surgery
* Patient undergoing psychological or psychiatric treatment
* Pregnant or breastfeeding woman, or a woman who is able to procreate without effective contraception
* Patient unable to follow the protocol as judged by the investigator
* Patient participating in another interventional research protocol involving a drug or medical device
* Patient under guardianship, curators or legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the relevance of the intervention of a physical therapist and a psychologist in the management of amputee patients in vascular surgery at 10 days post-operatively. | at 10 days post-operatively
  Mobility" and "Emotional Reactions" scores collected from the Nottingham Health Profile (NHP) scale at 10 days post-operatively
  It is a self-questionnaire for measuring perceived health in the general population or in patients. It allows the measurement of health-related quality of life. It is in the form of a questionnaire with 38 questions to which the patient must answer "yes" or "no". A score of 1 point will be awarded for a positive answer and 0 points for a negative answer.
  A score between 0 and 100 is thus obtained for each patient for each item. This percentage corresponds to the degree of difficulty perceived by the subject in the area of each of the headings.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie CORDON, Principal Investigator — Departmental Hospital Centre - Vendee
Locations (1):
- Departmental Hospital Centre - Vendee, La Roche-sur-Yon, France

REFERENCES:
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273